CLINICAL TRIAL: NCT05403021
Title: Piloting GETCare: A Remote Goal-based Education and Skills Training Program for Caregivers Poststroke
Acronym: GETCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Utah Occupational Therapy Association (Unknown)
Responsible Party: Principal Investigator, Jackie Einerson, Principal Investigator, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00129713; 00112906 (Other: IRB)
Record Dates: First submitted 2022-05-01; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Stroke
Keywords: caregiver; intervention; pilot; education; goals; skills
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: single-arm mixed method pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GETCare Intervention (Experimental)
  Interventions: Behavioral: GETCare Intervention

INTERVENTIONS:
Behavioral: GETCare Intervention — This 5-week intervention was administered remotely and individually to caregivers utilizing phone, email, and a secure online platform. The GETCare program was mostly self-led and included five weekly module education topics: basics of stroke, caregiver skills, caregiver changes, meaningful participation, and community resources. Each module incorporated (1) individualized education, (2) goal setting, (3) skills training, and (4) community resource recommendations. The program was led by a licensed occupational therapist who is a certified stroke rehabilitation specialist. The occupational therapist conducted weekly check-ins via email or phone focused on answering questions, tracking goal progress, and assisting in problem solving.

SUMMARY:
The purpose of this study was to evaluate the GETCare program, a Goal-based Education and skills Training program for Caregivers poststroke.

DETAILED DESCRIPTION:
The purpose of this study was to utilize a single-arm mixed method pilot trial to evaluate the5-week GETCare program with the following study aims: (1) explore feasibility and acceptability, (2) assess knowledge acquisition and goal attainment, and (3) test preliminary effects on key caregiver outcomes. This remote program included guided goal setting, individualized resource recommendations, and education modules.

ELIGIBILITY:
Inclusion Criteria:

* self-identification as a primary caregiver (direct care involvement) of someone who had a stroke (no restriction on stroke duration)
* ≥ 18 years old
* access to internet/telephone throughout the study
* able to speak, read, and understand English
* person with stroke expected to discharge within 1 month if still in the hospital

Exclusion Criteria:

* unable to read and follow basic instructions
* indicated the individual with stroke had no deficits poststroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | Baseline
  Scores range 0-40, higher score indicates higher perceived stress
Perceived Stress Scale | Post-intervention (approximately 6 weeks)
  Scores range 0-40, higher score indicates higher perceived stress
Revised Scale for Caregiving Self-efficacy | Baseline
  Scores range 0-100, higher score indicates higher self-efficacy
Revised Scale for Caregiving Self-efficacy | Post-intervention (approximately 6 weeks)
  Scores range 0-100, higher score indicates higher self-efficacy

SECONDARY OUTCOMES:
Modified Caregiver Strain Index | Baseline
  Scores range 0-26, higher score indicates higher caregiver strain
Modified Caregiver Strain Index | Post-intervention (approximately 6 weeks)
  Scores range 0-26, higher score indicates higher caregiver strain
Patient-Reported Outcomes Measurement Information System-43 Profile v2.1 | Baseline
  43 items across seven domains: physical function, anxiety, fatigue, depression, sleep disturbance, ability to participate in social roles and activities, and pain interference;
  Scores range 6-30 for each subscale. For subscales of anxiety, depression, fatigue, and sleep disturbance, higher scores indicate worse symptoms. For subscale of social participation, higher scores indicate improved symptoms. Subscales of physical function and pain interference were not included in analyses, since they were not expected to change through this intervention.
Patient-Reported Outcomes Measurement Information System-43 Profile v2.1 | Post-intervention (approximately 6 weeks)
  43 items across seven domains: physical function, anxiety, fatigue, depression, sleep disturbance, ability to participate in social roles and activities, and pain interference;
  Scores range 6-30 for each subscale. For subscales of anxiety, depression, fatigue, and sleep disturbance, higher scores indicate worse symptoms. For subscale of social participation, higher scores indicate improved symptoms. Subscales of physical function and pain interference were not included in analyses, since they were not expected to change through this intervention.
Neuro-Quality of Life (Neuro-QOL) Positive Affect and Well-being v1.0 | Baseline
  9 items; Scores range 9-45, higher score indicates higher positive affect and well-being
Neuro-Quality of Life (Neuro-QOL) Positive Affect and Well-being | Post-intervention (approximately 6 weeks)
  9 items; Scores range 9-45, higher score indicates higher positive affect and well-being
Knowledge assessment | Baseline
  Evaluate knowledge acquisition of weekly education topics; Scores range 0-35, higher score indicates higher knowledge
Knowledge assessment | Post-intervention (approximately 6 weeks)
  Evaluate knowledge acquisition of weekly education topics; Scores range 0-35, higher score indicates higher knowledge
Canadian Occupational Performance Measure | Baseline
  Assesses importance of goal, current performance of goal, and satisfaction with current performance of goal; Scores range 0-10, higher score indicates higher importance, performance, and satisfaction with performance
Canadian Occupational Performance Measure | Post-intervention (approximately 6 weeks)
  Assesses importance of goal, current performance of goal, and satisfaction with current performance of goal; Scores range 0-10, higher score indicates higher importance, performance, and satisfaction with performance

OTHER OUTCOMES:
Feedback survey | Post-intervention (approximately 6 weeks)
  Included a variety of questions (no/yes, Likert scales, and open-ended questions) regarding feedback of the intervention. For example, "Please indicate how helpful the additional handouts and videos were for you" (0 = not at all helpful, 1 = a little helpful, 2 = somewhat helpful, 3 = quite helpful, 4 = extremely helpful).

CONTACTS AND LOCATIONS:
Overall Officials: Jackie Einerson, MOT, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Einerson, J., & Terrill, A. (2019). GETCare: Development of a Comprehensive Education and Training Program For Care-Partners Post-Stroke. Archives of Physical Medicine and Rehabilitation, 100(10), e8. https://doi.org/https://doi.org/10.1016/j.apmr.2019.08.012